CLINICAL TRIAL: NCT01392612
Title: The Effect of Erythropoietin on Platelet Activation Markers: a Prospective Study in Healthy Volunteers
Brief Title: Erythropoietin and Platelet Activation Markers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Department of Clinical Pharmacology, Medical University of Vienna
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: EPO1
Record Dates: First submitted 2011-07-08; First posted 2011-07-12 (Estimated); Last update posted 2011-07-14 (Estimated); Status verified 2011-07

CONDITIONS: Thrombosis; Hypertension
Keywords: thrombosis; hypertension; gender; endothelium
MeSH Terms: conditions — Thrombosis; Hypertension; Coitus | interventions — Erythropoietin; Eosinophil Peroxidase

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Erythropoietin (Other): all subjects received epo iv.
  Interventions: Drug: erythropoietin

INTERVENTIONS:
Drug: erythropoietin — Subjects received one single intravenous injection of epoetin alpha (Erypo®, rhEPO, Ortho Biotech/Division of Janssen-Cilag Ag, Bridgewater, New Jersey, US) at a dose of 300 Units per kg bodyweight. Blood was sampled at baseline and 4, 24, 48 and 72 hours after administration of rhEPO during a biosimilarity trial.
  Other Names: epo

SUMMARY:
We hypothesized that the effect of erythropoietin may be reflected by changes in thromboxane B2 (TXB2) and endothelial cell function.

Six male and six female subjects received recombinant human epoetin alpha (Erypo®) intravenously (300 Units per kg). Biomarker levels were assessed at baseline and 4, 24, 48 and 72 hours after administration.

DETAILED DESCRIPTION:
Introduction: Erythropoietin (EPO) enhances formation of red blood cells and also affects thrombopoiesis and platelet function. We hypothesized that the effect of erythropoietin may be reflected by changes in thromboxane B2 (TXB2) and endothelial cell function.

Methods: Six male and six female subjects received recombinant human epoetin alpha (Erypo®) intravenously (300 Units per kg). Biomarker levels were assessed at baseline and 4, 24, 48 and 72 hours after administration.

Results: Epoetin alpha increased TXB2 levels, which reached significance at 48h (2.5- fold increase: 6.6±5ng/mL vs. 15±9ng/mL; p=0.044) and remained at that level at 72h. In line, epoetin alpha increased E-selectin levels by 25% already at 24h (39±21ng/ml vs. 49±26ng/ml; p<0.001) and stayed at this level until 72h (p<0.001). The raise in platelet activation markers corresponded with a 2-fold increase in reticulocyte count (81±17G/L vs. 43±10G/L; p<0.001) and a 9% increase in platelet count at 72h (224±45G/L vs. 244±52G/L; p=0.005). Thrombomodulin and von Willebrand factor concentrations were not significantly altered by epoetin alpha. Interestingly, gender differences in the baseline levels of E-selectin and thrombomodulin were observed. E-selectin and thrombomodulin levels were doubled in men compared to women (51±24ng/mL and 28±10ng/mL; p=0.025 and 30±5ng/mL vs. 16±5ng/mL; p=0.002, respectively).

Conclusion: Epoetin alpha increases levels of platelet activation markers. Further studies are needed to investigate whether measurement of TXB2 or E-selectin levels might be useful for estimation of thromboembolic risk during EPO-therapy.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female volunteers.
* Age between 18-40 years.
* Body mass index 17-27.
* Normal haemoglobin levels (Hb males 13.5-18g/dL, females 12-16g/dL).
* Reticulocyte count within reference values (32-110G/L).
* S-Iron within reference values (males 60-150µg/dl, females 40-150µg/dL).
* Serum ferritin within reference values (females 10-140µg/L, males 20-280µg/L).
* CRP within reference values (<1,0mg/dL).
* Signed informed consent.
* Normal findings in medical history and physical examination unless the investigator considers an abnormality to be clinically irrelevant for this study.
* Woman of child bearing potential must agree to practice effective barrier methods for birth control.

Exclusion Criteria:

* Smoking.
* Regular use of medication and food supplements containing iron.
* Abuse of alcoholic beverages and drugs.
* Participation in a clinical trial in the 3 weeks preceding the study.
* Foreseen inability to attend to scheduled study visits.
* Deficiency in folate (<3.4nmol/L) or vitamin B12 (<118pmol/L) (reevaluation after supplementation is allowed).
* Evidence of hypertension, pathologic hyperglycemia, hyperlipidemia. AST and/or ALAT > 3xULN (AST males > 105U/L, females >93U/; ALAT males > 135U/L, females >102U/L).
* Symptoms of a clinically relevant illness during 3 weeks prior the first study day.
* History or presence of gastrointestinal, liver or kidney disease, or other conditions known to interfere with distribution, metabolism or excretion of erythropoietin.
* Blood donation during the previous 3 weeks prior to the first study day.
* History of hypersensitivity erythropoietin.
* Pregnancy or lactation period.
* Any medical condition that, in the opinion of the investigator, would interfere with safety of the subject or interference of the objectives of the study.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2006-11; Primary Completion 2007-02 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
change in platelet activation markers | platelet activation markers were measured 4, 24, 48 and 72 hours after administration of iv EPO
  We wanted to examine whether levels of platelet activation markers change after administration of EPO and if they do, in which time frame it happens.

SECONDARY OUTCOMES:
change in erythropoietin levels | erythropoietin levels were measured 4, 24, 48 and 72 hours after administration
  We wanted to examine erythropoietin-levels after administration of EPO at mentioned time points.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Wolzt, Prof., Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria

REFERENCES:
- [Derived] Heinisch BB, Vcelar B, Kapiotis S, Blann A, Wolzt M, Siller-Matula JM, Jilma B. The effect of erythropoietin on platelet and endothelial activation markers: a prospective trial in healthy volunteers. Platelets. 2012;23(5):352-8. doi: 10.3109/09537104.2011.631621. Epub 2011 Nov 18. PMID 22098110